CLINICAL TRIAL: NCT00774995
Title: Study to Evaluate the Immune Response of Healthy Subjects Who Received Neonatal Vaccination Course With GSK Biologicals' Engerix™-B Vaccine, Approximately 20 Years Ago.
Brief Title: Immune Response of Healthy Subjects Who Received Neonatal Vaccination Course With Engerix™-B Vaccine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110073
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Engerix-B; Hepatitis B
MeSH Terms: conditions — Hepatitis B

ARMS (4):
- Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) (Experimental): Subjects who previously received HBV vaccine at 0, 1, 6 and 60 months (4 doses) and HBIg concomitantly at Month 0, and received a challenge dose of HBV vaccine after approximately 20 years (noted as Day 0) in the current study.
  Interventions: Biological: EngerixTM-B
- Engerix(3-dose)+HBIg (Experimental): Subjects who previously received HBV vaccine at 0, 1, 6 months (3 doses) and HBIg concomitantly at Month 0, and received a challenge dose of HBV vaccine after approximately 20 years (noted as Day 0) in the current study.
  Interventions: Biological: EngerixTM-B
- Engerix(4-dose) (Experimental): Subjects who previously received HBV vaccine at 0, 1, 6 and 60 months (4 doses) and received a challenge dose of HBV vaccine after approximately 20 years (noted as Day 0) in the current study.
  Interventions: Biological: EngerixTM-B
- Engerix(3-dose) (Experimental): Subjects who previously received HBV vaccine at 0, 1, 6 months (3 doses) and received a challenge dose of HBV vaccine after approximately 20 years (noted as Day 0) in the current study.
  Interventions: Biological: EngerixTM-B

INTERVENTIONS:
Biological: EngerixTM-B — Intramuscular injection, one dose.

SUMMARY:
This study will evaluate the immune response of healthy subjects who received neonatal vaccination course with GSK Biologicals' Engerix™-B vaccine, approximately 20 years ago. The presence of immune memory against hepatitis B surface antigen (HBsAg) in these subjects will be investigated by the administration of a challenge dose of hepatitis B vaccine and the comparison of their antibody concentration before and one month after vaccination.

This protocol posting deals with objectives & outcome measures of the booster phase. No new subjects will be recruited during this booster phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female who received the complete neonatal primary vaccination course of Engerix™-B in the 103860/273 primary study approximately 20 years earlier.
* Anti-HBs antibody concentrations less than the specified value at the last available follow-up time-point.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential,or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the Engerix™-B challenge dose, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressant or other immune-modifying drugs within six months prior to challenge dose administration.
* Planned administration/ administration of a vaccine not foreseen by the study protocol starting from 30 days before the challenge dose and ending 30 days after.
* Administration of a hepatitis B vaccine outside the context of this study between the follow-up time-point at which anti-HBs antibody concentrations was less than the specified value and the current challenge dose study visit.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the challenge dose visit or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Leroux-Roels G, Crasta PD, Hardt K. Persistence and immune memory to hepatitis B vaccine 20 years after primary vaccination of Thai infants, born to HBsAg and HBeAg positive mothers. Hum Vaccin Immunother. 2012 Jul;8(7):896-904. doi: 10.4161/hv.19989. Epub 2012 Jul 1. PMID 22777097
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Started | 9 | 16 | 8 | 16
Completed | 9 | 16 | 7 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose) | Total
Number analyzed (Participants) | 9 | 16 | 8 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.3 (0.5) | 19.6 (0.5) | 19.8 (0.46) | 19.5 (0.52) | 19.5 (0.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 7 | 21
  Male | 3 | 10 | 6 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Anamnestic Response to a Challenge Dose of Hepatitis B Virus (HBV) Vaccine as Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Description: Anamnestic response to the challenge dose is defined as: - At least (i.e. greater than or equal to) a 4-fold rise in post-challenge anti-HBsAg antibody concentrations in subjects seropositive at the last available follow-up time-point. -Post-challenge dose anti-HBsAg antibody concentrations >= 10 mIU/mL in subjects seronegative at the last available follow-up time-point.
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received the challenge dose of HBV vaccine and for whom data concerning immunogenicity measures were available at the post-HBV vaccine challenge dose time point.
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 8 | 14 | 6 | 15
Subjects | 8 | 13 | 6 | 14

2. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface (HBs) Antibody Concentrations Above Cut-off Values as Measured by ELISA.
Description: Cut-off values assessed were as follows: ≥3.3 milli-international units/milliliter (mIU/mL), ≥10 mIU/mL, ≥100 mIU/mL
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 8 | 14 | 6 | 15
Subjects
  ≥ 3.3 mIU/mL | 8 | 14 | 6 | 15
  ≥ 10 mIU/mL | 8 | 13 | 6 | 15
  ≥ 100 mIU/mL | 8 | 8 | 6 | 12

3. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface (HBs) Antibody Concentrations Above Cut-off Values as Measured by CLIA.
Description: Cut-off values assessed were as follows: ≥6.2 milli-international units/milliliter (mIU/mL), ≥10 mIU/mL, ≥100 mIU/mL
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 7 | 14 | 6 | 15
Subjects
  ≥ 6.2 mIU/mL | 7 | 12 | 6 | 15
  ≥ 10 mIU/mL | 7 | 12 | 6 | 15
  ≥ 100 mIU/mL | 7 | 7 | 6 | 11

4. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration as Measured by ELISA.
Description: Concentrations given as GMC expressed as milli-international unit per millilitre (mIU/mL).
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 8 | 14 | 6 | 15
mIU/mL | 2852.1 [1189.7 to 6837.3] | 163.8 [42.8 to 625.9] | 1420.2 [331.1 to 6090.9] | 515.5 [173.7 to 1530.3]

5. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration as Measured by CLIA.
Description: Concentrations given as GMC expressed as milli-international unit per millilitre (mIU/mL).
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 7 | 14 | 6 | 15
mIU/mL | 1831.6 [582.5 to 5758.9] | 165.6 [45.5 to 602.4] | 1335.2 [263.0 to 6779.0] | 454.1 [165.0 to 1250.0]

6. Primary Outcome: Number of Subjects With an Anamnestic Response to a Challenge Dose of Hepatitis B Virus (HBV) Vaccine as Measured by ChemiLuminescence ImmunoAssay (CLIA).
Description: as for outcome 1
Time Frame: One month after the hepatitis B vaccine challenge dose.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 7 | 14 | 5 | 12
Subjects | 7 | 11 | 5 | 12

7. Secondary Outcome: Number of Subjects Experiencing Any, Grade 3 and Related to Vaccination Unsolicited Symptoms.
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 symptom is any event that prevented normal activities. Related symptom is an event that was considered by investigator as causally related to the study vaccination.
Time Frame: During the 31-day follow-up period after the hepatitis B vaccine challenge dose.
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 9 | 16 | 8 | 16
Subjects
  Subjects with any symptoms | 1 | 0 | 0 | 0
  Subjects with grade 3 symptoms | 0 | 0 | 0 | 0
  Subjects with related symptoms | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects That Experienced Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period after the challenge dose (1 month).
Measure: Number; unit: Subjects
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Number analyzed (Participants) | 9 | 16 | 8 | 16
Subjects | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events: During the entire study period i.e. from Day 0 to Month 1; Unsolicited adverse events: During the 31 days (Day 0 to Day 30) post challenge dose.
Arm/Group | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) | Engerix(3-dose)+HBIg | Engerix(4-dose) | Engerix(3-dose)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/16 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 1/9 | 0/16 | 0/8 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix(4-dose)+HepatitisB(HB) Immunoglobulin (Ig) (N=9) | Engerix(3-dose)+HBIg (N=16) | Engerix(4-dose) (N=8) | Engerix(3-dose) (N=16)
Pyrexia (General disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL).The table shows updated results following complete retesting and reanalysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.